CLINICAL TRIAL: NCT01970098
Title: A Phase III Confirmatory Study of KPS-0373 in Patients With Spinocerebellar Degeneration (SCD)
Brief Title: A Confirmatory Study of KPS-0373 in Patients With Spinocerebellar Degeneration (SCD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KPS1301
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Spinocerebellar Degeneration
Keywords: Spinocerebellar degeneration (SCD); Thyrotropin-Releasing Hormone (TRH); Spinocerebellar Ataxia (SCA); Cortical Cerebellar Atrophy (CCA)
MeSH Terms: conditions — Spinocerebellar Degenerations; Spinocerebellar Ataxias

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- KPS-0373 (Experimental)
  Interventions: Drug: KPS-0373, High dose; Drug: KPS-0373, Low dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KPS-0373, High dose — 28 weeks
  Arms: KPS-0373
Drug: KPS-0373, Low dose — 28 weeks
  Arms: KPS-0373
Drug: Placebo — 28 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the superiority of KPS-0373 to placebo, and evaluate the safety and pharmacokinetics of KPS-0373 in SCD patients.

ELIGIBILITY:
Inclusion Criteria:

* Japanese SCD patients with mild to moderate ataxia

Exclusion Criteria:

* Patients with secondary ataxia
* Patients with clinically significant hepatic, renal, or cardiovascular dysfunction

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2013-10-09 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
SARA (Scale for the Assessment and Rating of Ataxia) | 24 weeks
  The change in the SARA total score at the time of final evaluation

SECONDARY OUTCOMES:
SF-8 (QOL) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuro Takei, Study Director
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Derived] Nishizawa M, Onodera O, Hirakawa A, Shimizu Y, Yamada M; Rovatirelin Study Group. Effect of rovatirelin in patients with cerebellar ataxia: two randomised double-blind placebo-controlled phase 3 trials. J Neurol Neurosurg Psychiatry. 2020 Mar;91(3):254-262. doi: 10.1136/jnnp-2019-322168. Epub 2020 Jan 14. PMID 31937586